CLINICAL TRIAL: NCT06173401
Title: A Randomized Phase III TriaL Comparing SingLe- Versus Multi-Fraction Spine STereotActic Radiosurgery for Patients With Spinal Metastases (ALL-STAR)
Brief Title: Comparing SingLe- Vs Multi-Fraction Spine STereotActic Radiosurgery in Spinal Metastases
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB-72248; BRN0060 (Other: OnCore number); NCI-2024-00695 (Registry Identifier: NCI- Clinical Trials Reporting Program)
Record Dates: First submitted 2023-11-28; First posted 2023-12-15 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Spinal Metastases
Keywords: spine stereotactic radiosurgery; cervical; lumbar; thoracic; metastases
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Single-fraction spine SRS (Experimental): Single-fraction spine SRS (22 Gy x 1)
  Interventions: Radiation: Single-fraction spine SRS
- Multi-fraction spine SRS (Experimental): Multi-fraction spine SRS (14 Gy x 2)
  Interventions: Radiation: Multi-fraction spine SRS

INTERVENTIONS:
Radiation: Single-fraction spine SRS — Treatment Arm 1: Single-fraction spine SRS (22 Gy x 1)
  Arms: Single-fraction spine SRS
Radiation: Multi-fraction spine SRS — Treatment Arm 2: Multi-fraction spine SRS (14 Gy x 2)
  Arms: Multi-fraction spine SRS

SUMMARY:
The goal of this study is to determine whether fractionated Stereotactic radiosurgery (SRS) for spine metastases is associated with improved local tumor control compared to single-fraction SRS. Patients will be randomized to treatment with spine SRS using either 22 Gy in 1 fraction or 28 Gy in 2 fractions.

ELIGIBILITY:
Inclusion Criteria:

* Histologically, cytologically, or radiographically confirmed diagnosis of metastatic cancer Age ≥ 18 years
* Patients who have cervical, thoracic, or lumbar spine metastasis that need treatment.
* Patients will have 1 to 3 separate spinal sites that require treatment.
* Each spinal site to be treated on trial will span 1-2 contiguous vertebral levels
* ECOG 0-2
* Negative serum or urine pregnancy test within 14 days prior to enrollment for people of childbearing potential or who are not postmenopausal
* people of childbearing potential and male participants who are sexually active must agree to use a medically effective means of birth control
* Ability to understand and the willingness to sign (personally or by a legal authorized representative) the written IRB approved informed consent document

Exclusion Criteria:

* Prior or planned radiation off study within or overlapping with study treatment site
* Inability to have either an MRI or a CT scan. Patients with pacemaker will be allowed to undergo CT instead of MRI
* Pediatric patients (age <18 years old), pregnant women, and nursing patients will be excluded
* Histology's of myeloma or lymphoma
* Patients with strength 1-3 (of 5), bladder incontinence, bowel incontinence, and/or bladder retention that is associated with spinal site to be treated
* Prior surgery to spinal site intended to be treated with protocol SRS
* Excluded those with SINS 13-18

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 274 (Estimated)
Dates: Start 2023-12-18 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Tumor control | 1 year
  To determine whether fractionated Stereotactic Radiosurgery (SRS) for spine metastases is associated with improved local tumor control at 1 year following SRS compared to single-fraction SRS.

SECONDARY OUTCOMES:
Euro-QOL EQ-5D-3L health-related quality of life questionnaire | 2 years
  To compare health-related quality of life (EQ-5D-3L) following SRS and assess patient-reported health related quality of life pertaining to mobility, self-care, usual activities, pain, and anxiety.
European Organization for Research and Treatment of Cancer (EORTC) QLQ-C30 health-related quality of life scale score | 2 years
  To compare health-related quality of life (EORTC QLQ-C30) following SRS and assess patient-reported health related quality of life pertaining to overall health and quality of daily life.
EORTC QLQ-BM22 health-related quality of life questionnaire | 2 years
  To compare health-related quality of life (EORTC QLQ-BM22) following SRS and assess patient-reported health related quality of life pertaining to pain associated with performing activities of daily life.
Pain Score | 1-2 weeks after SRS and 1, 3, 6, 12, 18, and 24 months following SRS
  Pain associated with the treated area will be assessed by asking patients to rate their pain on a 0-10 scale ("no pain" to "pain as bad as you can imagine")
Medication Intake | 1-2 weeks after SRS and 1, 3, 6, 12, 18, and 24 months following SRS
  Collect medications taken within the last 24 hours.
Number of participants with CTCAE grade grade 2 or higher adverse effects | 1 year
  To determine 1-year rate CTCAE grade 2 or higher adverse effects, following SRS
Rate of vertebral compression fracture | 1 year
  To determine 1-year rate of vertebral compression fracture (VCF), following SRS
Rate of local failure | 2 years
  To determine 2-year rate of local failure following SRS

CONTACTS AND LOCATIONS:
Overall Officials: Erqi Pollom, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Palo Alto, California, United States